CLINICAL TRIAL: NCT05362864
Title: Post-Market Clinical Follow-up Study on the ZNN™ Bactiguard ® Cephalomedullary Nails (Implants and Instrumentation). A Multicenter, Prospective, Consecutive Series
Brief Title: ZNN Bactiguard Cephalomedullary Nails PMCF Study
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CME2021-39T
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Osteotomy; Trochanteric Fractures; Sub-trochanteric Fractures; Femoral Shaft Fracture
Keywords: Bactiguard
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ZNN Bactiguard CMN: Subjects that have received or will receive the ZNN Bacitugard Cephalomedullaryl Nail to treat trochanteric, sub-trochanteric, and shaft fractures and osteotomies according to the cleared/approved indications.
  Interventions: Procedure: Fracture fixation via Intramedullary Nailing

INTERVENTIONS:
Procedure: Fracture fixation via Intramedullary Nailing — Fixation of trochanteric, sub-trochanteric, and shaft fractures and osteotomies.

SUMMARY:
This is a multicenter, prospective, Post-market Clinical Follow-up (PMCF) Study on the ZNN Bactiguard Cephalomedullary Nails. The objective of this study is to collect data confirming the safety, performance, and clinical benefit of the study device and instrumentation when used for the temporary internal fixation and stabilization of trochanteric, sub-trochanteric or shaft femoral fractures and osteotomies.

This is a CE-marked device already available on the market and the aim of the study is to comply with the post-market surveillance requirements.

DETAILED DESCRIPTION:
This study is a multicentre, prospective, post-market clinical follow-up study on the Zimmer Natural Nail (ZNN) Bactiguard Cephalomedullary Nails. The primary endpoint for this study is the assessment of performance by analyzing fracture/osteotomy healing within 12 months after fracture fixation. Radiological fracture healing is defined as bridging callus on at least three of the four cortices on the AP and lateral radiographs and clinically as full weight-bearing without pain.

The secondary endpoint is the assessment of safety, clinical benefit, and postop fracture-related infection (FRI). Safety will be evaluated by recording and analyzing the incidence and frequency of complications and adverse events. Relation of the events to implant, instrumentation and/or procedure should be specified. Clinical benefit will be assessed by recording patient-reported outcome measures (PROMs). FRIs will be classified according to the updated diagnostic algorithm defined by the FRI Consensus Group. Data will be collected at 6 weeks, 3 months, 6 months and 1 year after fracture fixation. The study will enroll patients implanted with the Zimmer Natural Nail Bactiguard Cephalomedullary Nail according to the approved/cleared indications. The sample size for this study is 150 study cases, and up to 10 sites in EMEA will participate.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older.
* Patient must have a signed EC approved informed consent.
* Patient must have a monolateral or bilateral trochanteric, sub-trochanteric, or shaft fracture requiring surgical intervention or osteotomy and be eligible for fixation by intramedullary nailing.
* Patient has been or is scheduled to be treated with the ZNN Bactiguard System Cephalomedullary Nail.
* Patient must be able and willing to complete the protocol required follow-up.
* Patients capable of understanding the surgeon's explanations and following his instructions.

Exclusion Criteria:

* Skeletally immature patients
* Medullary canal obliterated by a previous fracture or tumor
* Bone shaft having excessive bow or a deformity
* Lack of bone substance or bone quality, which makes stable seating of the implant impossible
* All concomitant diseases that can impair the operation, functioning or the success of the implant
* Insufficient blood circulation
* Infection
* Patient is unwilling or unable to give consent.
* Patient is a vulnerable subject (prisoner, mentally incompetent or unable to understand what participation to the study entails, subject with alcohol/drug addiction, known to be pregnant or breastfeeding).
* Patient anticipated to be non-compliant and/or likely to have problems complying with the follow-up program (e.g. patient with no fixed address, long-distance, plans to move during course of study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive series of patients aged 18 or older with femur fractures or osteotomies implanted with the ZNN Cephalomedullary Nail according to the approved/cleared indications.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Performance of the study device by analyzing fracture/osteotomy healing at 12 months after fracture fixation. | 12 months after fracture fixation
  Performance will be assessed by analyzing fracture/osteotomy healing at 12 months after fracture fixation. Fracture healing will be assessed clinically and radiologically:
  * Radiological fracture healing is defined as bridging callus on at least three of the four cortices on the AP. and lateral radiographs
  * Clinical fracture healing is defined as full weight-bearing without pain.

SECONDARY OUTCOMES:
Safety assessment by recording and analyzing incidence and frequency of adverse events. | 6 weeks and 3, 6, and 12 months after fracture fixation
  Recording and analyzing incidence and frequency of adverse events.
Oxford Hip Score | 3, 6, and 12 months after fracture fixation
  Patient-Reported Outcome Measures (PROMs) that document hip function and pain. It's used as a surrogate to assess function and pain of the operated limb.
EQ-5D Health Questionnaire | 3, 6, and 12 months after fracture fixation
  Patient-reported outcome completed by the patient. It assesses the general health status of the patient and it can be used to derive a quality of life index used for health economics considerations.
Rate of fracture-related infections | 6 weeks and 3, 6, and 12 months after fracture fixation
  Fracture-related infections are diagnosed in accordance with the algorithm described in M McNally, G Govaert, M Dudareva, M Morgenstern, W J Metsemakers, EFORT Open Rev 2020;5:614-619.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Rohmer, Study Director — Zimmer Biomet
Locations (3):
- Centre Hospitalier de Douai, Douai, France, France
- Spain (2):
  - Hospital Rio Hortega, Valladolid, Castille-La Mancha
  - Hospital Clinico de Valencia, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No